CLINICAL TRIAL: NCT07188714
Title: Preoperative Prediction of VATS Strategy in Parapneumonic Effusion
Brief Title: Video-assisted Thoracoscopic Surgery (VATS) Has Revolutionised Management of Complicated PPE, Our Study to Determine VATS Decortication Technique is Needed, Compared to VATS Debridement in PPE, Also RAPID Score and Pleural US Parameters Can Predict Which VATS Procedure is Needed.
Acronym: VATs-PPE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hamed Farrag Qenawy, assistant lecturer, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VATs,Assiut University 1
Record Dates: First submitted 2025-09-03; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Parapneumonic Effussion
Keywords: VATs in Parapneumonic effussion

STUDY DESIGN:
Intervention Model Description: Patients with complicated pleural infections, who don't improve after antibiotics and drainage of fluid by chest tube, will undergo surgery. The procedure may be debridement, where the surgeon only removes pus and debris, wash the thoracic cavity with saline and inserts chest tube. If the surgeon finds it necessary, he will proceed to decortication, where he also peels-off the thick infected pleura covering the lung to allow lung regain its size and help improvement. Follow up will include, clinical assessment, laboratory tests, periodic CXR to decide whether it's appropriate to remove the chest tube or not
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- decortication arm (Active Comparator): patients with PPE complicated by stage 3 empyema will underwent decortication technique
  Interventions: Procedure: VATs decortication
- debridement arm (Active Comparator): patients with PPE complicated by stage 2 empyema will underwent debridment technique
  Interventions: Procedure: VATs debridement

INTERVENTIONS:
Procedure: VATs decortication — A long thoracoscopic instruments are to be used for dissection, evacuation of pus and removal of the visceral peel at the surface of the lung. Instruments will be introduced below the lens in cases of uniportal procedure. Two ports VATS will be used early in this series by adding another 3-4 cm incision in the 3rd or 4th intercostal space anterior axillary line, scope will be introduced through the lower port and instruments will be introduced through the other.
  Irrigation with warm saline is to be done; breaking up the fine adhesions, the surgeon will take off the thick visceral peel over the lung surface, opening the fissures using combination of blunt and sharp dissection leaving the parietal pleura.
  Arms: decortication arm
Procedure: VATs debridement — Removal of pus, debris, granulation tissue is to remove as much as possible of the empyema biofilm while freeing the lung from any loculations.
  Following debridement and flushing the pleural cavity by warm saline, the attending anaesthiologist is to modify the ventilatory settings to attain the maximally allowed degree of lung expansion (TV criteria/peak/plateau/PV curve). Then, instillation of saline to obliterate the pleural cavity until saline leaks back from the operating port. If leakage starts after instillation of ≤200 cc. (obliteration of the whole pleural cavity including the cost phrenic angle will be assumed, lung is to be considered sufficiently expanded, and VATS will be withheld at debridement step. On the other hand, if leakage starts after instillation of ≥ 200 cc, lung entrapment and failure of expansion will be assumed, and surgery will proceed to VATS decortication to achieve reasonable lung expansion
  Arms: debridement arm

SUMMARY:
Video-assisted thoracoscopic surgery (VATS) has revolutionised management of complicated parapneumonic effusion ( PPE). So our study is prospective cohort study will be conducted at Departments of Chest Diseases and Cardiothoracic Surgery, Assiut University Hospitals

* Aims: to determine the frequency of which VATS technique is needed (decortication versus debridement ) and to verify whether baseline RAPID score and pleural US parameters can predict which VATS procedure (decortication vs. debridement) in patients with complicated PPE will need, upon intra-operative exploration to compare the time to ICT removal after lung expansion and length of hospital stay in patients with PPE undergoing VATS via either debridement or decortication approach .
* Subjects: All patients with PPE presenting with suggestive symptoms,signs or radiological studies which display compatible patterns of PPE:

  1. Inclusion criteria:

     1. Age > 18 years
     2. Patients diagnosed with PPE who are confirmed by (aspiration of frank pus from pleural cavity, positive culture for bacterial infection, pleural fluid with a pH ⩽7.2 (measured by blood gas analyser), low glucose level (⩽3 mmol/L or ⩽55 mg•dL-1), lactate dehydrogenase (LDH) >200 IU/L) in a patient with clinical evidence of infection .
     3. Failed resolution of parapneumonic effusion.
  2. Exclusion criteria:

     1. Patients unfit for/ or declining surgical intervention.
     2. Iatrogenic or traumatic pyothorax.
     3. Haemothorax or chylothorax regardless the etiology.
     4. Exudative pleural effusion due to medical conditions other than pneumonia .
* Sample size was calculated using Epi-info software version 7.2.5.0. The total sample size needed to detect such an estimate with 95% confidence level and 10% margin of error will be 95 patients
* Research outcome measures:

  1. Primary (main):

     * Number of the patients who will receive either VATS technique (and the respective percentage in relation to the total patients)
     * Preoperative Adjusted RAPID score and US findings (fluid volume, echogenicity, pleural thickening, consolidation and other incidental findings).
     * Assessment the radiological signs of lung expansion

CXR/US scores:

* Failure: Chest X-ray scoring 0 and chest US scoring 0.
* Partially successful: Chest X-ray scoring 1 or 2 and chest US scoring 1.
* Successful: Chest X-ray scoring 3 or 4, and chest US scoring 2 or 3.

B. Secondary (subsidiary):

* Time to ICT removal (days). ICT tube will be removed based on the MDT joint decision according to the patients' individual course. Tube removal is contemplated upon clinical resolution, complete fluid drainage, full lung expansion and absence of pleural air in CXR, in the absence of air leak, chest ultrasound to assess if there is residual pleural effusion.
* Length of Hospital Stay (days)
* Status at discharge (ICT removed or not)
* Patients reported outcomes:

  * Postoperative pain (VAS) at discharge time
  * Resumption of usual activities (self-care routine with assistance - unassisted self-care- other activities indoors- independent indoors and outdoors activities) by attending the patient to the hospital within 30 days post discharge.
  * Mortality rate within 30 days postoperative.

DETAILED DESCRIPTION:
* Type of the study: Prospective Cohort Study.
* Study Group: VATS debridement versus VATS decortication.
* Study Setting: Departments of Chest Diseases and Cardiothoracic Surgery, Assiut University Hospitals.
* Study subjects:

All patients with PPE presenting with suggestive symptoms (acute onset fever, cough, expectoration ± pleuritic chest pain or hemoptysis), signs (fever, increased TVF, Bronchial breath sound, localized crepitation) or radiological studies (CXR and pleural US ±CT Chest) which display compatible patterns (semihomgenous opacity with blunting of the costophrenic angle, homogenous opacity suggestive loculated effusion, air bronchogram):

1. Inclusion criteria:

   1. Age > 18 years
   2. Patients diagnosed with PPE who are confirmed by (aspiration of frank pus from pleural cavity, positive culture for bacterial infection, pleural fluid with a pH ⩽7.2 (measured by blood gas analyzer), low glucose level (⩽3 mole/L or ⩽55 mg•dL-1), lactate dehydrogenase (LDH) >200 IU/L) in a patient with clinical evidence of infection .
   3. Failed resolution of parapneumonic effusion:
2. Exclusion criteria:

   1. Patients unfit for/ or declining surgical intervention.
   2. Iatrogenic or traumatic pyothorax.
   3. Haemothorax or chylothorax regardless the aetiology.
   4. Exudative pleural effusion due to medical conditions other than pneumonia (suspected or proven Para malignant effusion, associated pulmonary embolism, autoimmune, pancreatic or esophageal disease, gynecological disorder, and drug-induced pleural effusion).
3. Sample Size Calculation:

   The sample size was calculated using Epi-info software version 7.2.5.0 . The total sample size needed to detect such an estimate with 95% confidence level and 10% margin of error will be 95 patients.

   -Study tools :all patients will be subjected to:
   1. Demographic data (age, gender) and clinical data (including comorbidities -such as underlying COPD, D.M, HTN, cardiac, hepatic, or renal diseases, immunodeficiency or administration of immunosuppressive therapy- symptoms and their duration, time to admission, time before ICT insertion and duration of antibiotics used) will be collected and documented.
   2. Laboratory testing:

      * Samples for baseline Complete blood count (CBC) with differential count, renal (serum urea and creatinine) and liver function tests (total protein, ALT, AST, albumin), coagulation profile (PT, PC, INR), LDH,ESR, and CRP will be , fasting and 2 hour postprandial blood sugar level will be collected, analyzed and their results will be documented.
      * Biochemical and microbial analysis of the pleural effusion will be conducted. This will include pleural pH, glucose level , LDH, total protein and albumin, culture and sensitivity for bacteria, as well as direct smear for A.F.B./Gene Expert (if pleural tuberculosis is suspected) by thoracentesis using ultrasound to guide selection of an adequate length needle. At least 10 mm depth to do diagnostic thoracentesis .
   3. Radiological studies before and after intervention:

      i) Chest X ray (CXR) PA/Lateral film. ii) Contrast-enhanced CT chest if deemed necessary by the MDT. Data about extent of the effusion, presence of loculi or pleural thickening, as well as the underlying lesions (pneumonia, mass, nodules) will be documented iii) Chest US:
      * The device:

      Curvilinear US probe (Samsung Madison CO-LTD.42 .Teheran-ro-108-gil.Gangnam-gu. Seoul. Korea) that generates a frequency range of 2-5 MHz which has great penetration but lower resolution .
      * Examination protocol:

      Patients are to be examined in the supine and sitting positions, arms raised and hands placed at the back of the head to expand the intercostal spaces and rotate the scapula outward. Examination will be performed systematically through the intercostal spaces in six vertical lines which are mid clavicular, anterior axillary, mid axillary, posterior axillary, mid scapular and paravertebral .and will cover 8 zones in each lung side (supra-mammary, mammary ,infra-mammary, upper axillary ,lower axillary ,supra-scapular ,inter-scapular , infrascapular ) .

      Sonographic Findings (include fluid volume, fluid echogenicity, pleural thickening, findings demonstrating the underlying pneumonia (hyperechoic comma-shape artifacts representing air bronchogram/C profile), other incidental findings (nodules, hypoechoic lesions).

      - Fluid volume: First, the maximal inter-pleural distance at posterior-lateral Alveolar and pleural syndrome (PLAPS) point is measured during expiration in a semi-recumbent position. Then, the volume of the pleural fluid will be calculated using Balik's Formula where .

      V(ml)= 20 x Distance (mm)

      - Echogenicity: Effusion is defined as anechoic when it is echo-free, as complex non-septate when echogenic material is inside the effusion, and as complex septate when floating fibrin strands or septa are found inside the effusions.
   4. Assessment of Mortality and Morbidity Risks:

      Adjusted RAPID score is a simple and easily calculated score that assesses mortality risk for patients with pleural infections. The score entails 8 parameters (Renal (urea), age, fluid purulence, infection source, dietary (albumin), diabetes mellitus, renal insufficiency (dialysis), immunosuppression are assigned . The total adjusted RAPID score (0-10 points) represents the sum of the points assigned to the 8 parameters together, on the basis of which the patient's risk for 90 days mortality is determined .
   5. Assessment of Fitness for Anesthesia and Surgery: ASA score (American Society of Anesthesiologists Physical Status ) It is a standardized way to assess a patient's overall health and fitness before surgery. It uses a scale of I to VI, with I being a healthy patient and VI being a deceased organ donor. An "E" is added to the number if the procedure is an emergency. According to age, diseases severity, associated comorbidities, the anaestheology team assign the patient into one of six classes that define the patient's fitness status in a descending rank.
   6. Anesthesia:

   The type of the anesthesia that will be administrated to the patient (general or regional) will be documented, as well as the drugs used during anesthesia as (inhalational anesthetics like sevoflurane, and intravenous agents like Propofol and remifentanil).

   7- VATS technique:

   • Materials :

   The following equipment is used to perform a VATS:

   1-5 or 10 mm high-resolution fiber-optic thoracoscopy with a 0° or 30° lens 2-A light source with a cable 3-Video monitors 4-Thoracoscopic instruments (scissors, hook or straight-blade cautery, biopsy forceps, grasper, and dissector) 5-Endoscopic stapler if resection is planned 6-Trocars 7-Thoracotomy tray (to convert to open procedure if needed) 8-Chest tubes and drainage devices 9-Sterile gloves, gowns, and drapes 10-Double-lumen endotracheal tube
   * Procedure steps :

     * The whole series will be operated upon under general anesthesia, using a double-lumen tube for selective ventilation.
     * Patients will be placed in a decubitus position on an operating table with a standby set of thoracotomy instruments ready in case of conversion.
     * A small incision (3-5 cm) is to be made in the 5th intercostal space anterior axillary line then dissection of the subcutaneous tissue and muscles was done. Port inserted with A 30-degree lens (Karl-Storz) in a 10-mm sheath thoracoscopy was introduced at the top of the incision.
     * After opening the port site, a gentle digital palpation to push the lung away from chest wall and create a space where camera can be introduced. Using the suction tip or a sponge on a stick afterward to further continue the dissection under vision .
   * Debridement technique :

   The aim of debridement (removal of pus, debris, granulation tissue) is to remove as much as possible of the empyema biofilm while freeing the lung from any loculations.

   Following debridement and flushing the pleural cavity by warm saline, the attending anaesthiologist is to modify the ventilatory settings to attain the maximally allowed degree of lung expansion (TV criteria/peak/plateau/PV curve). Then, instillation of saline to obliterate the pleural cavity until saline leaks back from the operating port. If leakage starts after instillation of ≤200 cc. (obliteration of the whole pleural cavity including the cost phrenic angle will be assumed, lung is to be considered sufficiently expanded, and VATS will be withheld at debridement step. On the other hand, if leakage starts after instillation of ≥ 200 cc, lung entrapment and failure of expansion will be assumed, and surgery will proceed to VATS decortication to achieve reasonable lung expansion.
   * Decortication technique :

     - For cases with lung entrapment by thick visceral peel or clotted hemothorax, irrigation with warm saline is to be done; breaking up the fine adhesions, the surgeon will take off the thick visceral peel over the lung surface, opening the fissures using combination of blunt and sharp dissection leaving the parietal pleura.

     - A long thoracoscopy instruments are to be used for dissection, evacuation of pus and removal of the visceral peel at the surface of the lung. Instruments will be introduced below the lens in cases of uniport procedure. Two ports VATS will be used early in this series by adding another 3-4 cm incision in the 3rd or 4th intercostal space anterior axillary line, scope will be introduced through the lower port and instruments will be introduced through the other.

     - After performing decortication, a warmed saline solution for flushing again inside the chest cavity through a 50-cc syringe for irrigation then suctioned after anesthetist start to ventilate this side and air leak was checked.

     -Decortication will be considered completed when near full lung expansion takes place with anesthetist inflating the lung with pressure between 30 and 35 mmHg. Failure to get the whole lung inflation needs a revision of the decortication and either continuing VATS or converting to open surgery depending on the comfort of the operator.

     8-Post-Operative Care:
   * ICT insertion :

     - Tools: 2 hemostats, nylon suture (0 or 0-1), scalpel size (11blade), suction apparatus, water seal drainage, chest tube ranges from 28-32 French for Para pneumonic effusion.
     * Chest tube will be inserted from the same port site then secured by sutures and other ports closed in standard fashion, so termination the surgical procedure and start recovery from anesthesia.
   * Recovery from anesthesia:

   Awaken a patient after general anesthesia by gradually reduce and eventually stop the anesthetic medications. The patient will then be monitored closely as they naturally wake up and regain consciousness, breathing on their own.

   • Site of admission: All Patients will be sent to the ward or the intermediate care unit, as a part of the institution's protocol.

   • Analgesia: According to pain ladder score :

   The original ladder mainly consisted of three steps:

   1-First Step: Mild pain: non-opioid analgesics such as non-steroidal anti-inflammatory drugs (NSAIDs) or acetaminophen with or without adjuvants.

   2-Second Step: Moderate pain: weak opioids (hydrocodone, codeine, tramadol) with or without non-opioid analgesics and with or without adjuvants.

   3-Third Step: Severe and persistent pain: potent opioids (morphine, methadone, fentanyl, oxycodone, buprenorphine, tapentadol, hydromorphone, oxymorphone) with or without non-opioid analgesics, and with or without adjuvant.

   Adjuvants, also called co-analgesics, include antidepressants, including tricyclic antidepressants (TCAs) such as amitriptyline and nortriptyline, serotonin-norepinephrine reuptake inhibitors (SNRIs) such as duloxetine and venlafaxine, anticonvulsants like gabapentin and pregabalin, topical anesthetics (e.g., lidocaine patch), topical therapies (e.g., capsaicin), corticosteroids, bisphosphonates, and cannabinoids .

   • Early mobilization and physiotherapy will be encouraged in all patients until discharge.

   9-Follow Up protocol postoperative: i) Amount of drained fluid daily in cc, color (serous, pus, blood or serosanguinous) (pre-operative and post-operative).

   ii) CXR and Chest US in day prior to surgery and 1 day postoperative then at discharge :

   • Chest X-ray is to be scored into: No change in the first X-ray before VATS takes score ( 0) Less than 1/3 improvement/lung expansion takes score(1). Improvement between 1/3 and 2/3 takes score (2). More than 2/3 improvement without complete clearance of effusion takes score(3).

   Complete radiological clearance/complete lung expansion takes score(4)
   * Chest US findings is to be scored into:

   No change takes score(0). Dissolution of adhesions in some regions takes score(1). Dissolution of adhesions in all regions with residual pleural affection takes score(2).

   Total adhesion dissolution without residual pleural lesion takes score(3). iii) Presence of air leak at discharge. iv) Visual analogue Sore (VAS): It is a scale from 0-10 cm with 0 value on the left side representing maximum comfort and 10 representing maximum discomfort on the right side will be assessed at in day prior to surgery and 1 day postoperative then at discharge .

   -Research outcome measures:

<!-- -->

1. Primary (main):

   * Number of the patients who will receive either VATS technique (and the respective percentage in relation to the total patients)
   * Preoperative Adjusted RAPID score and US findings (fluid volume, echogenicity, pleural thickening, consolidation and other incidental findings).
   * Assessment the radiological signs of lung expansion:

   CXR/US scores:

   -Failure: Chest X-ray scoring 0 and chest US scoring 0.
   * Partially successful: Chest X-ray scoring 1 or 2 and chest US scoring 1.
   * Successful: Chest X-ray scoring 3 or 4, and chest US scoring 2 or 3.

   B. Secondary (subsidiary):

   • Time to ICT removal (days): ICT tube will be removed based on the MDT joint decision according to the patients' individual course. Tube removal is contemplated upon clinical resolution, complete fluid drainage, full lung expansion and absence of pleural air in CXR, in the absence of air leak, chest ultrasound to assess if there is residual pleural effusion.
   * Length of Hospital Stay (days)
   * Status at discharge (ICT removed or not)
   * Patients reported outcomes:

     * Postoperative pain (VAS) at discharge time
     * Mobility (bed bound- need for assistance as wheelchair or help of relatives to move -freely and independently ambulatory) by attending the patient to the hospital within 30 days post discharge.
     * Resumption of usual activities (self-care routine with assistance - unassisted self-care- other activities indoors- independent indoors and outdoors activities) by attending the patient to the hospital within 30 days post discharge.
     * Mortality rate within 30 days postoperative, documentation of the cause of death will be attempted.
   * Complication : minor as bleeding, wound infection, surgical emphysema, postoperative blood transfusion or major as worsening of pneumonia, sepsis, persistent air leak, need to re-exploration.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Patients diagnosed with PPE who are confirmed by (aspiration of frank pus from pleural cavity, positive culture for bacterial infection, pleural fluid with a pH ⩽7.2 (measured by blood gas analyser), low glucose level (⩽3 mmol/L or ⩽55 mg•dL-1), lactate dehydrogenase (LDH) >200 IU/L) in a patient with clinical evidence of infection [6].
3. Failed resolution of parapneumonic effusion:

Given a patient-to-patient variability in response to medical treatment, therapeutic pleurocentesis and ICT drainage, a MDT involving consultant cardiothoracic surgeons and consultant pulmonologist are to discuss enrolled cases individually , reach consensus, and declare failure of medical treatment or ICT drainage and need for surgical intervention , based on combination of clinical , laboratory, and radiological parameters (persistence of fever. Elevated Wbcs, respiratory symptoms, pleural fluid loculi inaccessible by ICT, lung entrapment despite complete drainage of fluid or large bronchopleural fistula

Exclusion Criteria:

1. Patients unfit for/ or declining surgical intervention.
2. Iatrogenic or traumatic pyothorax.
3. Haemothorax or chylothorax regardless the aetiology.
4. Exudative pleural effusion due to medical conditions other than pneumonia (suspected or proven Para malignant effusion, associated pulmonary embolism, autoimmune, pancreatic or oesophageal disease, gynaecological disorder, and drug-induced pleural effusion).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2025-10-25 (Estimated); Primary Completion 2027-09-10 (Estimated); Study Completion 2028-02-10 (Estimated)

PRIMARY OUTCOMES:
Assessment the radiological signs of lung expansion | perioperative
  CXR/US scores:
  * Failure: Chest X-ray scoring 0 and chest US scoring 0.
  * Partially successful: Chest X-ray scoring 1 or 2 and chest US scoring 1.
  * Successful: Chest X-ray scoring 3 or 4, and chest US scoring 2 or 3.
Preoperative Adjusted RAPID score and US findings | the baseline
  Preoperative Adjusted RAPID score which determine what is the technique will be used ( decortication or debridement ) as shown :
  Adjusted RAPID score is a simple and easily calculated score that assesses mortality risk for patients with pleural infections. The score entails 8 parameters (Renal (urea), age, fluid purulence, infection source, dietary (albumin), diabetes mellitus, renal insufficiency (dialysis), immunosuppression are assigned as seen in Figure(1). The total adjusted RAPID score (0-10 points) represents the sum of the points assigned to the 8 parameters together, on the basis of which the patient's risk for 90 days mortality is determined .
  Risk categories :
  score 0-2 low risk score 3-4 intermediate risk score 5-7 high risk score 8-10 very high risk

SECONDARY OUTCOMES:
Time to ICT removal (days) | through study completion, an average of 30 days
  ICT tube will be removed based on the MDT joint decision according to the patients' individual course. Tube removal is contemplated upon clinical resolution, complete fluid drainage, full lung expansion and absence of pleural air in CXR, in the absence of air leak, chest ultrasound to assess if there is residual pleural effusion.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Mohamed Hashem, MD, Study Chair — Assiut Medical School; Hend Mohamed Sayed, MD, Study Chair — Assiut Medical School
Locations (1):
- Assiut university- Faculty of medicine, Asyut, Assiut Governate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bernstein WK, Deshpande S. Preoperative evaluation for thoracic surgery. Semin Cardiothorac Vasc Anesth. 2008 Jun;12(2):109-21. doi: 10.1177/1089253208319868. PMID 18635562
- [Background] Chambers A, Routledge T, Dunning J, Scarci M. Is video-assisted thoracoscopic surgical decortication superior to open surgery in the management of adults with primary empyema? Interact Cardiovasc Thorac Surg. 2010 Aug;11(2):171-7. doi: 10.1510/icvts.2010.240408. Epub 2010 May 3. PMID 20439299
- [Background] Towe CW, Carr SR, Donahue JM, Burrows WM, Perry Y, Kim S, Kosinski A, Linden PA. Morbidity and 30-day mortality after decortication for parapneumonic empyema and pleural effusion among patients in the Society of Thoracic Surgeons' General Thoracic Surgery Database. J Thorac Cardiovasc Surg. 2019 Mar;157(3):1288-1297.e4. doi: 10.1016/j.jtcvs.2018.10.157. Epub 2018 Nov 28. PMID 33198004
- [Background] Dean NC, Griffith PP, Sorensen JS, McCauley L, Jones BE, Lee YC. Pleural Effusions at First ED Encounter Predict Worse Clinical Outcomes in Patients With Pneumonia. Chest. 2016 Jun;149(6):1509-15. doi: 10.1016/j.chest.2015.12.027. Epub 2016 Jan 16. PMID 26836918
- See also: Related Info — http://www.pubmed.gov/